CLINICAL TRIAL: NCT00654966
Title: Evaluation of the Effects of Urotensin-II and Soluble Epoxide Hydrolase Inhibitors on Skin Microvessel Tone in Patients With Heart Failure, and in Healthy Volunteers.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Monash University (Other)
Responsible Party: Prof Henry Krum, Monash University / Alfred Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CP-02/08; 77/08
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Heart Failure
Keywords: Urotensin II; Soluble epoxide hydrolase; Iontophoresis; Healthy volunteers
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Heart failure patients
  Interventions: Drug: Urotensine II; Drug: Soluble epoxide hydrolase
- 2 (Active Comparator): Healthy subjects
  Interventions: Drug: Urotensine II; Drug: Soluble epoxide hydrolase

INTERVENTIONS:
Drug: Urotensine II — A few drops of the drug will be administered to the skin by iontophoresis.
Drug: Soluble epoxide hydrolase — A few drops of the drug will be administered to the skin by iontophoresis.

SUMMARY:
Urotensin II (U-II) is newly discovered protein that may play an important role in human health and disease. U-II has been found to be a potent vasoconstrictor (narrower of blood vessels) which therefore may be involved in important diseases such as chronic heart failure - CHF (weak heart muscle disease). Many vasoconstrictors have been found to have effects on key organs such as the heart. Preliminary data by our group have demonstrated this is true of U-II. Recent evidence shows that in CHF, U-II levels in the blood are increased.

The proposed study seek to determine the effect of blocking a possible downstream mediator of U-II on blood vessels by administration of soluble epoxide hydrolase inhibitor (sEHI). There will be 2 study groups 1) Healthy volunteers and, 2) CHF patients.

Each arm of the study will run independently and will require 16 participants each (16 normal subjects and 16 CHF subjects). Participants will be screened to ensure that they are eligible. CHF patients will be required to withdraw from their CHF medication 24 hours prior to the study day (except for diuretics). On the study day, sEHI will be administered on the skin of participants in 3 asceding dosages. The technique to be used is iontophoresis. This is a non invasive technique in which a small amount of the compound is placed on the skin of the forearm. The drug is delivered across the skin by passing a small electric current over the area. The change in blood flow is then measured and analysed. We will also administer U-II agonist, noradrenaline, and distilled water (all via iontophoresis). Noradrenaline will be used a positive constrictor control. Change in blood flow will be assessed by Laser Doppler Velocimetry.

If it is found that the sEHI is able to prevent blood vessel constriction in CHF patients, then it may represent a major therapeutic advance in the management of CHF.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed written informed consent.
* Male/Female over 18 and under 80 years of age.
* Females must be non-pregnant, non-lactating and using reliable means of contraception (surgical sterilisation or a barrier method such as a condom). The oral contraceptive pill is an exclusion to this study.
* Patients with CHF will be required to have left ventricular fractional shortening [LVFS] of <22% or LVEF < 40% and New York Heart Association functional class [NYHA FC] II-III symptoms
* Body mass index (BMI) between 18-35 kg/m2.
* Screening clinical laboratory tests including liver function tests and HbA1c are within the normal reference range for the investigative site.
* Electrocardiogram (ECG) results considered within normal limits, as determined by the Investigator.

Exclusion Criteria:

* Smokers
* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, neurological, or other disorders capable of altering the absorption, metabolism, or elimination of drugs, or of constituting a risk factor when exposed to the study medication.
* Those requiring concomitant medications that will affect cardiovascular or endothelial function or blood pressure control (eg cholesterol lowering medication, hormone replacement therapy, aspirin, NSAIDS).
* Patients receiving Hormone Replacement Therapy.
* Known allergy or hypersensitivity to urotensin or urotensin receptor antagonists or its excipients, or related drugs, or a history of relevant adverse drug reactions of any origin.
* Regular alcohol intake greater than 14 units/week or is unwilling to comply with the alcohol prohibition for the duration of the study (1 unit of alcohol is equivalent to: 12 ounces of beer, 4 ounces of wine, or 1 ounce of 50-proof hard liquor).
* History of drug abuse.
* Screening biochemistry > 20 % outside normal limits.
* Patients who are thought to be terminally ill or immuno-compromised
* Patients who have previously been enrolled in this study or have received other experimental medications in the last 4 weeks.
* Patients who are unlikely to comply with study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To compare the vasoactive role of Soluble epoxide hydrolase in the healthy subjects and CHF patients with iontophoresis. | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Henry Krum, MBBS FRACP PhD, Principal Investigator — Monash University / Alfred Hospital
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia